CLINICAL TRIAL: NCT00123448
Title: Mirroring a Movement
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050205; 05-N-0205
Record Dates: First submitted 2005-07-21; First posted 2005-07-22 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-07-02

CONDITIONS: Healthy
Keywords: Mirror Neurons; fMRI; Premotor Cortex; gesture; Healthy Volunteer; HV
MeSH Terms: conditions — Gestures

SUMMARY:
This study will determine if the type of gesture, increased quantity of an image, and the number of times a face is shown repeating a gesture bring about activation in the "mirror neurons." Researchers aim to learn about which areas of the brain are necessary to perform certain cognitive tasks-that is, relating to a person's thinking or remembering-especially visual and motor tasks. Because one way humans learn is by imitation, a mechanism is required to transfer the behavior the person adopts from others through observation. This type of learning could be based on a mechanism similar to that provided by mirror neurons. From previous studies it has been learned that the observation of hands and mouths has brought about the most effective ways of activating the mirror neurons.

Patients ages 21 to 55 who are in good health, are right handed, are not pregnant, and are native speakers of English may be eligible for this study. There will be about 24 participants.

Patients will undergo a magnetic resonance imaging (MRI) scan. Before the scan, they will complete a safety questionnaire about the presence of any metal in their bodies. Patients are at risk for injury from the MRI magnet if they have pacemakers, dental implants or other devices. Female patients will undergo a pregnancy test. The technique MRI uses includes a strong magnetic field and radio waves to obtain images of body organs and tissues. During the initial MRI scan, patients will lie still on a table that will slide into the enclosed tunnel of the scanner. They will be in the scanner for about an hour. During the procedure, they may be asked to lie as still as possible for up to 20 minutes at a time. As the scanner takes pictures, patients will hear knocking or beeping sounds. Each participant will wear earplugs to reduce this noise. They will be able to communicate with the MRI staff at all times during the scan, and they may ask to be removed from the machine at any time. The functional MRI (fMRI) scan will involve taking pictures of the brain while patients are performing tasks. All the tasks will be explained, and patients will have the chance to practice them before entering the scanner. During the fMRI, patients will view short film segments of people making gestures. Before and after the scan, patients will be asked to complete several short questionnaires. The testing sessions will take a total of about 2 hours.

Participants will receive compensation for their time and inconvenience, with a maximum payment of $200. This study will not have a direct benefit for participants.

DETAILED DESCRIPTION:
Objective: The purpose of the protocol is to determine the effects of the social content of gestures on brain activation patterns. We will localize the extent and areas of brain activation by using functional MRI during observation of gesture varied by type of gesture, number of images shown at a time, and number of times a subject is exposed to a face.

Study Population: Healthy, normal adult volunteers will participate in a gesture observation experiment using functional magnetic resonance imaging (fMRI).

Design: The experiment we are conducting will employ an event-related design to determine whether increasing the social content of the gesture spreads activation from traditional sensorimotor regions engaged in mirror movement activity to regions in the prefrontal cortex (PFC) concerned with processing social behavior.

Outcome Measures: The data collected will consist of accuracy measures of cognitive performance, fMRI images, and post-questionnaire results. The results gained from this protocol will provide evidence for a social effect of gesturing.

ELIGIBILITY:
* INCLUSION CRITERIA:

In all the studies, subjects will consist of healthy, native English-speaking, right-handed volunteers, as measured by the Edinburgh Handedness Inventory. Subjects will range in age from 21 to 55 years old and they will be included regardless of race or gender.

EXCLUSION CRITERIA:

Non-native English speakers and non-right handers will be excluded as mentioned above, as will non-neurologically normal volunteers. Subjects younger than 21 and older than 55 will be excluded. A urine pregnancy test will be employed with all women of childbearing age. The results must be negative in order to proceed with the MRI.

Subjects with any of the following: aneurysm clip; implanted neural stimulator; implanted cardiac pacemaker or auto-defibrillator; cochlear implant; ocular foreign body, e.g. metal shavings; permanent eyeliner; insulin pump; or irremovable body piercing will be excluded from the study due to the possible dangerous effects of the magnet upon metal objects in the body. Subjects taking central nervous system active medications will be excluded.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36
Dates: Start 2005-07-20; Study Completion 2008-07-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Belliveau JW, Rosen BR, Kantor HL, Rzedzian RR, Kennedy DN, McKinstry RC, Vevea JM, Cohen MS, Pykett IL, Brady TJ. Functional cerebral imaging by susceptibility-contrast NMR. Magn Reson Med. 1990 Jun;14(3):538-46. doi: 10.1002/mrm.1910140311. PMID 2355835